CLINICAL TRIAL: NCT03829540
Title: A Phase I, Multicenter Study of CD4- Directed Chimeric Antigen Receptor Engineered T-cells (CD4CAR) in Patients With Relapsed or Refractory CD4+ Hematological Malignancies
Brief Title: CD4CAR for CD4+ Leukemia and Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huda Salman (Other)
Collaborators: iCell Gene Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Huda Salman, Director, Brown Center for Immunotherapy, Don Brown Professor of Immunotherapy, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-ICG122-101; FD-R-006820-01 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2018-12-19; First posted 2019-02-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: T-cell Lymphoma; T-cell Leukemia
Keywords: CD4; T-cell; lymphoma; leukemia; chimeric antigen; CAR-T
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, T-Cell; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Redirected autologous T cells transduced with the anti-CD4 lentiviral vector (referred to as "CD4CAR" cells)
  Interventions: Biological: CD4CAR

INTERVENTIONS:
Biological: CD4CAR — CD4CAR cells transduced with a lentiviral vector to express the single-chain variable fragment (scFv) nucleotide sequence of the anti-CD4 molecule derived from humanized monoclonal ibalizumab and the intracellular domains of CD28 and 4-1BB co-activators fused to the CD3ζ T-cell activation signaling domain administered by IV infusions as a single dose

SUMMARY:
This study is designed as a single arm open label Phase I, 3x3, multicenter study of CD4-directed chimeric antigen receptor engineered T-cells (CD4CAR) in patients with relapsed or refractory T-cell leukemia and lymphoma. Specifically, the study will evaluate the safety and feasibility of CD4CAR T-cells. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
The study will be performed as a dose-escalation protocol. Due to the relatively low incidence and prevalence of cluster of differentiation 4-positive (CD4+) hematological malignancies and the associated aggressive nature of these diseases and the sequel of treatment failure, the investigators expect to recruit 20 subjects at Stony Brook, Indiana University, and other identified sites with an expected dropout rate of 25% primarily due to rapid progression or death and screen and or manufacturing failure. Taking this into account, the investigators expect to treat 15 patients. The study will utilize autologous CD4CAR T-cells that are engineered to express a chimeric antigen receptor (CAR) targeting CD4 that is linked to the cluster of differentiation 28 (CD28), 4-1BB, cluster of differentiation 3-zeta (CD3ζ) signaling chains (third generation CAR).

At entry, disease status will be staged and investigators will determine if the subject has adequate T cell number for apheresis and for manufacturing CD4CAR cells. Qualifying subjects will be leukapheresed to obtain large numbers of peripheral blood mononuclear cells (PBMC) for the manufacturing. Next, participants will receive conditioning chemotherapy. If tumor burden is sufficiently reduced (screening step), participants will receive CD4CAR cells by infusion on Day 0 of treatment.

For cell harvest, 12-15-liter apheresis procedure will be performed at the apheresis center with the intention to harvest at least 50x10^9-nucleated cells to manufacture CD4CAR T-cells. A portion of the pheresed cells will also be cryopreserved for FDA look-back requirements and for further research. The T-cells will be purified from the PBMC, transduced with CD4CAR lentiviral vector, expanded in vitro, and then frozen for administration. Each dose will be stored in either one or two bags. The route of administration is by IV infusion and the duration of infusion will be approximately 20 minutes. Each bag will contain an aliquot (30-50 mL) of liquid suitable for freezing, and containing the following infusible grade reagents (% v/v): 4.5% human serum albumin with 10% DMSO. The cell product is expected to be ready for release approximately 3-4 weeks after apheresis.

If the disease progresses during the manufacturing period participants may be excluded from the study. Minimal chemotherapy to keep the disease under control in the meanwhile is allowed if deemed necessary by investigators.

A single dose of CD4CAR transduced T cells will consist of the cell number for the dose level to be infused.

Post-infusion monitoring of CD4CAR T-cells: Subjects will have blood drawn for cytokine levels, CD4CAR Transgene Copy Number (PCR) and flow cytometry in order to evaluate the presence of CD4CAR cells on days 0, 1, 3, 5, 7, 14, 28, and 42 following infusion (or as clinically needed). Cytokines levels will be evaluated per schedule above in addition to and as needed every 8 +/- 2 hours as feasible if/when CRS occurs and until resolution. Active monitoring of fungal and viral infections during treatment while utilizing standard prophylaxis recommended for HIV-positive patients with T-cell aplasia and those undergoing allogeneic stem cell transplant. Investigators plan to collect data about clinicoradiologic measurements of residual tumor burden starting on day 6 and weekly afterward until day 42 and then monthly for 6 months. This will be followed by quarterly clinical evaluations for the next two (2) years with a medical history, physical examination, and comprehensive blood testing. After these short- and intermediate-term evaluations are performed, these patients will enter a rollover study to assess for disease-free survival (DFS), relapse, and the development of other health problems or malignancies where follow-up will be up tp twice a year by phone and a questionnaire for an additional thirteen (13) years. The treating physician will decide to proceed with allogeneic or autologous transplant when needed.

Dose of CD4CAR description: the main objective of this study is to establish a recommended dose and/or schedule of CD4CAR. The guiding principle for dose escalation in phase I is to avoid unnecessary exposure of patients to sub-therapeutic doses (i.e., to treat as many patients as possible within the therapeutic dose range) while preserving safety and maintaining rapid accrual. Investigators will use the rule-based traditional Phase I "3+3" design for the evaluation of safety. Based on lab experience in mice the starting dose (dose level 1) for the first cohort of three patients in phase I portion of the study will be 8x10^5 cells. The dose escalation or de-escalation will follow a modified Fibonacci sequence as below.

If more than one patient out of the first cohort of three patients in dose level 1 experience dose limiting toxicity (DLT), the trial will be placed on hold. If zero or one out of three patients in the first cohort of dose level 1 experience DLT, three more patients will be enrolled at dose level 1; the dose escalation continues until at least two patients among a cohort of six patients experience DLT (i.e., ≥33% of patients with a DLT at this dose level)

* If one of the first three patients in dose level 1 experiences a DLT, three more patients will be treated at dose level 1.
* If none of the three patients or only one of the 6 patients in the dose level 1 experiences a DLT, the dose escalation continues to the dose level 2
* If one of the first three patients in dose level 2 experience a DLT, three more patients will be treated at dose level 2
* If none of the three patients or only one of the 6 patients in the dose level2 experiences a DLT, the dose escalation continues to the dose level 3
* If one of the first three patients in dose level 3 experiences a DLT, three more patients will be treated at dose level 3
* If none of the three patients or only one of the 6 patients in the dose level 3 experiences a DLT, dose level 3 will be declared the maximum tolerated dose (MTD) and will be used as the recommended phase II dose (RP2D) for the phase II portion of the study.

In summary, the dose escalation continues until at least two patients among a cohort of six patients experience DLT (i.e., ≥33% of patients with a DLT at that dose level). The recommended dose for phase II trials is defined as one dose level below this toxic dose level. Since some grade 3 and possibly 4 toxicities are highly likely to be reversible, grade 3 infectious, hematological and vascular toxicities will not be considered DLTs mandating dose reduction. Also allergic or infusion-related reactions ≤ grade 3 will not be counted as DLTs. There will be no intra-patient dose escalation or reduction.

To allow for full spectrum toxicity duration evaluation and reporting, no patients within the same or a different cohort will be initiated on lymphodepleting chemotherapy sooner than 42 days from the initiation date of the preceding patient.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, an individual will be enrolled if they meet the following criteria:

1. Patients must voluntarily sign and date informed consent forms that state his or her willingness to comply with all study procedures and availability for the duration of the study.
2. Age 12 years old or older
3. Subjects with any documented CD4+ T cell hematologic malignancies. Male and female subjects with CD4+ T-cell hematologic malignancies with either relapsed or refractory disease (including those patients who have undergone a prior transplant (if allogeneic, subjects are eligible if there are no remaining donor cells) and patients with an inadequate response after 4-6 cycles of standard chemotherapy) are eligible. Response criteria for each disease subset will be evaluated based on Standard of Care Guidelines.
4. Creatinine clearance of > 60 ml/min (or otherwise non clinically-significant, per study investigator)
5. ALT/AST < 3 x ULN
6. Bilirubin < 2 x ULN
7. No supplemental oxygen at rest Note: Pulmonary Function Test (PFT) only required per treating physician discretion
8. Adequate cardiac function with EF of ≥50%
9. Adequate venous access for apheresis and no other contraindications for leukapheresis

Exclusion Criteria

1. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential (see definition below) must have a negative serum or urine pregnancy test prior to initiation of conditioning chemotherapy, per research sites' clinical policy.
2. Uncontrolled active infection necessitating systemic therapy.
3. Active hepatitis B or hepatitis C infection. Active hepatitis C is defined as the hepatitis C antibody is positive while quantitative HCV RNA results exceed the lower detection limit.

   Note the following subjects will be eligible:
   * Subjects with a history of hepatitis B but have received antiviral therapy and have nondetectable viral DNA for 6 months prior to enrollment are eligible
   * Subjects seropositive for HBS antibodies due to hepatitis B virus vaccine with no signs or active infection (Negative HBs Ag, HBc and HBe Ags) are eligible
   * Subjects who had hepatitis C but have received antiviral therapy and show no detectable hepatitis C virus (HCV) viral RNA for 6 months are eligible
   * If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
4. Concurrent use of systemic glucocorticoids in greater than replacement doses (unless as a part of a standard of care salvage therapy or conditioning protocol), or steroid dependency defined in rheumatological and pulmonary diseases as uninterrupted corticosteroid intake for more than a year at a dosage of 0.3 mg/kg/day or greater, and where the underlying disease worsens on temporary stoppage of steroid therapy, with symptoms of steroids withdrawal (eg, lethargy, headache, weakness, pseudorheumatism, emotional disturbances, etc) precipitated by the temporary stoppage.

   Subjects who receive daily corticosteroids in replacement doses can be included in the study. The replacement doses are defined as following:
   1. Hydrocortisone 25mg/day or less
   2. Prednisone 10mg/day or less
   3. Dexamethasone 4mg or less Note: Recent or current use of inhaled glucocorticoids is not exclusionary, as this route pertains extremely minimal systemic penetration.
5. Any uncontrolled active medical disorder that would preclude participation as outlined in the opinion of the treating investigator and/or study chair
6. HIV infection.
7. Subjects declining to consent for treatment
8. Subjects who have received or will receive live vaccines within 30 days before the first experimental cell treatment. Inactivated seasonal flu vaccination is allowed.
9. Subjects with active autoimmune diseases who need systematic treatments (such as disease modifying agents, corticosteroids and immunosuppressive drugs) in the last 2 years. Note: Replacement therapy (thyroxine, insulin or physiological corticosteroid replacement therapy (up to10 mg of oral daily prednisone or equivalent in hydrocortisone and dexamethasone) to treat adrenal dysfunction or pituitary dysfunction) is not considered as systematic therapy. Subjects who need inhalation corticosteroid therapy can be included in this trial. Subjects with vitiligo or in long-term remission of pediatric asthma or allergic diseases can be included in this trial.
10. Subjects with a history of mental disorders or drug abuse that may influence treatment compliance.
11. Active malignancy not related to a T-cell malignancy that has required therapy in the last 3 years or is not in complete remission. Exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy. Other similar malignant conditions may be discussed with and permitted by the Principal Investigator.
12. Treatment with any investigational cell/gene therapy within the past 6 months
13. Treatment with any investigational anticancer agent within 14 days of study entry or 5 half-lives (whichever is shorter)

Eligibility for Conditioning Chemotherapy

1. Specific organ function criteria for cardiac, renal, and liver function must be similar to initial inclusion values.
2. Review of co-morbidities to confirm no major changes in health status (examples of major changes include heart attack, stroke, and any major trauma).
3. Planned infusion dose was successfully manufactured and met release criteria.
4. Negative pregnancy testing (if applicable).

Eligibility for CD4CAR infusion:

Inclusion

1. Afebrile and not receiving antipyretics, and no evidence of active infection.
2. Specific organ function criteria for cardiac, renal, and liver function must be similar to initial inclusion values. The following test does not need repeated: EF if obtained within 6 weeks of initial assessment.
3. If previous history of corticosteroid chemotherapy, subject must be off all but adrenal replacement doses 3 days before the CD4CAR infusion.

Exclusion

Note: A subject may still receive the CD4CAR infusion up to 10 days post conditioning chemotherapy as long as they do not meet any of the following at time of infusion:

1. Requirement for supplemental oxygen to keep saturation greater than 95% or presence of radiographic abnormalities on a clinically indicated chest x-ray that are progressive.
2. New cardiac arrhythmia not controlled with medical management.
3. Hypotension requiring pressor support.
4. Positive blood cultures for bacteria, fungus, or virus within 48-hours of T cell infusion.

Contraception and Reproductive Potential Guidelines Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test prior to conditioning chemotherapy.

Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception from time of consent through at least 90 days after CD4CAR infusion.

Acceptable birth control includes a combination of two of the following methods:

* Condoms (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormonal-based contraception Subjects who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy, salpingotomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception. Acceptable documentation of sterilization, azoospermia, and menopause is specified next:

Written or oral documentation communicated by clinician or clinician's staff of one of the following:

* Physician report/letter
* Operative report or other source documentation in the subject record (a laboratory report of azoospermia is required to document successful vasectomy)
* Discharge summary
* Laboratory report of azoospermia
* Follicle stimulating hormone measurement elevated into the menopausal range

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2041-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 18-24 months
  To assess the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD4 lentiviral vector (referred to as "CD4CAR" cells) according to CTCAE grading. The feasibility of treating those adverse events and their duration till resolution will also be described.

SECONDARY OUTCOMES:
Duration of in vivo survival of the CD4CAR. | 18-24 months
  Persistence of CD4CAR will be monitored by measuring the CD4CAR transgene copy number at variable time points.
Rate of manufacturing failure | 18-24 months
  The number of failed manufacturing attempts of CD4 CAR, per subject and overall, in this patient population. Manufacturing failure is defined as failure to manufacture the adequate CD4CAR cell dose for the particular cohort the patient is enrolled on. Three manufacturing attempts per patient are allowed.
Clinical Response | 18-24 months
  Clinical response to T-cell infusion will be evaluated by comparing disease before and after infusion identified by:
  * standard imaging (PET CT or PET MRI) for lymphoma patients
  * bone marrow biopsy for leukemia patients
  * peripheral blood cells morphology, flow cytometry panel, immunohistochemistry, and other blood molecular markers for both lymphoma and leukemia.
Trafficking of CD4CAR at tumor sites and at sites with significant toxicity | 18-24 months
  Quantification of both of CD4CAR by research flow cytometry and transgene copy number by polymerase chain reaction (PCR) will be measured at tumor sites in bone marrow and lymph nodes at variable time points if applicable. Same tests will be done on biopsies of organs that shows significant toxicity if need be.
Number of participants with immune reactions against CD4CAR | 18-24 months
  The absolute and relative number of subjects who develop immune reactions against the treatment over a period of 2 years. Human anti-mouse antibody (HAMA) ELISA tests will be carried out in the blood of participants at multiple times after initial treatment.
Serum cytokines levels | 18-24 months
  Serum cytokine levels will be evaluated on Day 2, 4, 7, 11, 14, 21, 28 in addition to planned monitoring during CRS approx. every 8 hours and until resolution. These cytokines include interleukin-6 (IL-6), interferon-γ, tumor necrosis factor, IL-2, IL-2-receptor-a, IL-8, and IL-10
Determine CD4CAR cell subsets during proliferation | 18-24 months
  Participants' blood will be tested by research flow cytometry to determine the relative abundance of cellular subsets that may result from CD4CAR T cells upon their proliferation. These subsets include Tcm, Tem, and Tregs, when feasible.
Overall survival and causes of death | throuh study completion (i.e.up to 15 years)
  Descriptive reporting on subjects survival duration post CAR infusion, and if they die, what is the cause of death
New onset malignancies post CD4CAR treatment | throuh study completion (i.e.up to 15 years)
  Descriptive reporting of any other cancers that may be diagnosed after enrollment in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Huda Salman, MD, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Albert Einstein Health Network, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No